CLINICAL TRIAL: NCT05092347
Title: A Dose Escalation and Proof-of-Concept Study of Vonsetamig (BCMA × CD3 Bispecific Antibody) for Desensitization of Chronic Kidney Disease Patients in Need of Kidney Transplantation Who Are Highly Sensitized to Human Leukocyte Antigen
Brief Title: A Study to Learn How Safe and Tolerable Vonsetamig is in Adult Patients With Chronic Kidney Disease (CKD) Who Need Kidney Transplantation and Are Highly Sensitized to Human Leukocyte Antigen (HLA)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5459-RT-1944
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: Kidney Transplant; Hemodialysis; Desensitization; Human Leukocyte Antigen (HLA)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vonsetamig (Experimental)
  Interventions: Drug: Vonsetamig

INTERVENTIONS:
Drug: Vonsetamig — Administered by intravenous (IV) infusion
  Other Names: BCMAxCD3; REGN5459

SUMMARY:
The purpose of this study is to determine whether vonsetamig will safely decrease anti-HLA antibodies to allow for kidney transplantation.

Vonsetamig is being studied for treatment of patients in need of kidney transplantation who are highly sensitized to HLA.

The study is looking at several other research questions, including:

* Side effects that may be experienced from taking vonsetamig
* How vonsetamig works in the body
* How much vonsetamig is present in the blood
* If vonsetamig works to lower levels of antibodies to HLA

ELIGIBILITY:
Key Inclusion Criteria:

1. Has Chronic Kidney Disease (CKD) requiring hemodialysis, and awaiting kidney transplant on the United Network for Organ Sharing (UNOS), with a cPRA ≥99.9%, or those with a cPRA >98% (98.1% to 99.8%) who have spent 5 years or longer on the waitlist, as defined in the protocol
2. Adequate hematologic and adequate hepatic function as defined in the protocol
3. Willing and able to comply with clinic visits and study-related procedures

Key Exclusion Criteria:

1. Current or active malignancy not in remission for at least 1 year
2. Central nervous system (CNS) pathology or history of CNS neurodegenerative or movement disorders
3. Patients who have had their spleen removed, including patients with functional asplenia
4. Patients who have received a stem cell transplantation within 5 years
5. Use of investigational agents within 8 weeks or 5 half-lives of study drug administration (whichever is larger)
6. Total plasma IgG <300 mg/dL at screening
7. Continuous systemic corticosteroid treatment with more than 10 mg per day of prednisone (or anti-inflammatory equivalent) within 72 hours of start of study drug administration
8. Received a calcineurin inhibitor (eg, tacrolimus, cyclosporine) within 30 days of study drug administration
9. Received cyclophosphamide, rituximab, obinutuzumab, other anti-CD20 or B cell-depleting agents, or proteasome inhibitors or anti-CD38 therapies (eg, isatuximab, daratumumab) within 12 months of study drug administration
10. Prior treatment with any anti-BCMA antibody (including antibody drug conjugate or bsAb) or BCMA-directed CAR-T cell therapy, as described in the protocol
11. Has received a COVID-19 vaccination, as described in the protocol

Note: Other protocol defined inclusion / exclusion criteria apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2026-03-24 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event(s) of interest (AEI) from the first dose through end of the safety observation period | Up to approximately 6 weeks
Incidence and severity of treatment-emergent adverse events (TEAE)s from the first study drug dose up to the end of the study | Up to 78 weeks
  TEAEs include adverse events of special interest (AESI) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Proportion of Participants with a clinically meaningful reduction in anti-HLA alloantibodies | Up to 78 weeks
  Clinically meaningful reduction in anti-HLA alloantibodies are defined as either:
  * Reduction in Calculated panel-reactive antibody (cPRA) from baseline, or
  * Reduction in the peak (immunodominant) anti-HLA mean fluorescence intensity (MFI) to <5,000, or by ≥50% by Single antigen bead (SAB) assay
Maximum reduction in the peak (immunodominant) MFI of anti-HLA alloantibodies from baseline | Up to 78 weeks
Percent change from baseline in the peak (immunodominant) MFI | Up to 78 weeks
Percent change from baseline in the sum of MFI of anti-HLA alloantibodies using the SAB assay | Up to 78 weeks
Time to first clinically meaningful reduction in anti-HLA alloantibody levels by SAB assay | Up to 78 weeks
  Defined as peak anti-HLA alloantibody MFI <5,000 or ≥50% reduction
Time to maximal reduction in anti-HLA alloantibody levels by SAB assay | Up to 78 weeks
  Defined as peak anti-HLA alloantibody MFI <5,000 or ≥50% reduction
Maximum reduction in cPRA from baseline | Up to 78 weeks
Time to first clinically meaningful reduction in cPRA | Up to 78 weeks
Time to maximal reduction in cPRA from baseline | Up to 78 weeks
Duration of a reduction in peak anti-HLA alloantibody to MFI <5,000 or by ≥50% by SAB assay | Up to 78 weeks
Duration of maximal reduction in anti-HLA alloantibody MFI by SAB assay | Up to 78 weeks
Duration of maximal reduction in cPRA by SAB assay | Up to 78 weeks
Serum concentration of Immunoglobulin (Ig) classes over time | Up to 78 weeks
Percent change from baseline of serum concentration of Ig classes | Up to 78 weeks
Concentration of vonsetamig in serum over time | Up to 78 weeks
Incidence of treatment-emergent anti-drug antibodies (ADAs) to vonsetamig over time | Up to 78 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (10):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine, Orange, California
  - Connie Frank Transplant Center at UCSF, San Francisco, California
  - Yale University of Medicine, New Haven, Connecticut
  - Medstar Georgetown Transplant Institute - 2-PHC, Washington D.C., District of Columbia
  - Comprehensive Transplant Center, Chicago, Illinois
  - John Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - New York University Langone Health, New York, New York
  - Penn Transplant Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/